CLINICAL TRIAL: NCT03125447
Title: Posture and Mobility Influence on Attention Capacity in Former Premature Children at 6 Years of Age.
Brief Title: Mobility and Attention Capacity in Former Premature Children
Acronym: PAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Jean-Michel HASCOET, Professor, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2017-A00327-46
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Attention Concentration Difficulty; Mobility Limitation
Keywords: Prematurely born children; Attention function; Posture; Mobility
MeSH Terms: conditions — Mobility Limitation | interventions — Calcium Carbonate

STUDY DESIGN:
Intervention Model Description: Attention capacity will be compared in three situations of posture/mobility in a group of prematurely born children, and compared to the same situations in a group of term born children
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prematurely born children (Experimental): Speed and accuracy answer to visual stimuli evaluated in 3 distinct posture/mobility situations
  Interventions: Other: speed and accuracy answer to visual stimuli
- Term born children (Active Comparator): Speed and accuracy answer to visual stimuli evaluated in 3 distinct posture/mobility situations
  Interventions: Other: speed and accuracy answer to visual stimuli

INTERVENTIONS:
Other: speed and accuracy answer to visual stimuli — A yellow fish swimming over a blue-green background will appear on the screen of virtual glasses. The child will have to give as fast as possible the direction of the fish pushing the left or right button of a computer mouse

SUMMARY:
Attention functions have a major impact on children's social and school behavior. They are an important issue for prematurely born children often seen as having learning difficulties and being restless, when it could be an adaptative answer to attention disorders. The aim of this study is to evaluate attention capacity in former premature children aged 6-7 years old with regards to different postures or mobility, for the attention functions of orienting, alerting and executive control. The Attention Network Test using reaction time and accuracy to visual stimuli will be used to evaluate attention functions in each posture and mobility.

DETAILED DESCRIPTION:
Attention functions have a major impact on children's social, school and emotional adjustment. They are one of the most common issues for prematurely born children with implications in academic and social-behavioral functioning. Prematurely born infants are often seen as having excessive mobility or being restless when it could be an adaptative answer to attention disorders leading to learning difficulties. Respecting spontaneous mobility could improve attention performance in vulnerable children. The aim of the study is to evaluate global attention performance of former premature children at the preschool age of 6 to 7 years. This evaluation will be done in three usual postures or mobility, and for the 3 attentional functions of orienting, alerting or executive control. They will be compared within the prematurely born children group and to term born controls of the same age. The Attention Network Test adapted to children by Rueda et al (Neuropsychologia 2004) using reaction time and accuracy to visual stimuli will be used to evaluate attention functions. Presentation of stimuli through virtual video glasses and collection of answers will be done thanks to a specific software.

ELIGIBILITY:
Main Inclusion Criteria:

* Children born before 35 weeks gestation and routinely followed for their prematurity in the follow-up clinic of the Maternite Regionale Universitaire

Healthy term born children recruited after information leaflet displayed in the University but not the Hospital

Main Exclusion Criteria:

* Children with a visual or motor disability preventing the realization of the test

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Reaction time to respond to visual stimuli appearance | 5 minutes
  48 trials of swimming fishes displayed for a maximum of 2500 msec in different conditions: the reaction time in msec will be recorded and evaluated

SECONDARY OUTCOMES:
Accuracy to the response to visual stimuli direction | 5 minutes
  48 trials of swimming fishes to the right or the left hand side where the child has to give the right direction of the fish

CONTACTS AND LOCATIONS:
Locations (1):
- Maternity Hospital CHRU, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rosenbaum J, Ceyte H, Hamon I, Deforge H, Hascoet AMJ, Caudron S, Hascoet JM. Influence of body mobility on attention networks in school-aged prematurely born children: A controlled trial. Front Pediatr. 2022 Sep 8;10:928541. doi: 10.3389/fped.2022.928541. eCollection 2022. PMID 36160773
- [Derived] Ceyte H, Rosenbaum J, Hamon I, Wirth M, Caudron S, Hascoet JM. Mobility may impact attention abilities in healthy term or prematurely born children at 7-years of age: protocol for an intervention controlled trial. BMC Pediatr. 2018 Aug 6;18(1):264. doi: 10.1186/s12887-018-1229-1. PMID 30081860